CLINICAL TRIAL: NCT03566082
Title: Post-Approval Study of the R3 Biolox Delta Ceramic Acetabular System - Europe
Acronym: R3 EU PAS
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Collaborators: eResearchTechnology, Inc (Industry); M Squared Associates, Inc. (Industry); ExecuPharm PAREXEL (Industry); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: R11019
Record Dates: First submitted 2018-01-10; First posted 2018-06-21 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-08

CONDITIONS: Degenerative Joint Disease of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post Approval Study: The PAS cohort consisted of 137 subjects who were implanted with the R3 delta Ceramic Acetabular System (DoD) in the pivotal study. These patients will continue to be followed to 10 years post-operatively.
  The primary endpoint for the PAS study is implant survivorship at 10 years post study procedure.

SUMMARY:
The purpose of this prospective, multicenter, single arm study is to confirm the long-term safety and effectiveness of the R3 delta Ceramic Acetabular System PMA (P150030) by evaluating long-term (10 years after surgery) follow-up results.

DETAILED DESCRIPTION:
This PAS is a long-term follow-up of the R3 delta Ceramic Acetabular System (DOD) hips enrolled in the study that was analyzed for the Premarket Approval Application (PMA) Study. The PMA Study analyzed 3 Year postoperative follow-up data on Biolox delta ceramic-on-Biolox delta ceramic (DOD) and Oxidized zirconium-on-Crosslinked Polyethylene (OxZr/XLPE) hips, enrolled and followed in a European Post-market Study ("A prospective, multicenter, non-randomized, clinical outcome study of the R3 Acetabular System in patients with degenerative hip disease").

The purpose of this prospective, multicenter, single arm study is to confirm the long-term safety and effectiveness of the R3 delta Ceramic Acetabular System PMA (P150030) by evaluating long-term (10 years after surgery) follow-up results. Hips are evaluated at the following intervals: 5, 7, 10 years postoperative. The primary study endpoint is implant survivorship at 10 years post surgery.

ELIGIBILITY:
Inclusion Criteria:

Patient is 18-75 years old and he/she is skeletally mature

* Patient requires primary total hip arthroplasty due to non-inflammatory degenerative joint disease (e.g. osteoarthritis, post-traumatic arthritis, avascular necrosis, dysplasia/ developmental dysplasia of the hip) or inflammatory joint disease (e.g., rheumatoid arthritis)
* Patient has met an acceptable preoperative medical clearance and is free from or treated for cardiac, pulmonary, hematological, etc., conditions that would pose excessive operative risk
* The patient is willing to comply the follow-up schedule

Exclusion Criteria:

Patient has active infection or sepsis (treated or untreated)

* Patient is a prisoner or has an emotional or neurological condition that would pre-empt their ability or unwillingness to participate in the study including mental illness, mental retardation, linguistic insufficiencies (i.e. immigrants), or drug/alcohol abuse,
* Patients with acute hip trauma (femoral neck fracture)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical study can fulfill its objectives only if appropriate subjects are enrolled. All relevant medical and non-medical conditions should be taken into consideration when deciding whether a particular patient is suitable.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2009-05-28 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- AZ Nikolaas, Sint-Niklaas, Belgium
- Finland (2):
  - HUS Peijaksen sairaala, Ortopedia ja traumatologia, Helsinki
  - TYKS Turku University Hospital, Turku
- La Paz Hospital, Madrid, Spain
- The Royal Orthopaedic Hospital, NHS Foundation Trust, Birmingham, United Kingdom

REFERENCES:
- [Derived] Davis ET, Remes V, Virolainen P, Gebuhr P, Van Backle B, Revell MP, Kopjar B. Mid-term outcomes of the R3 delta ceramic acetabular system in total hip arthroplasty. J Orthop Surg Res. 2021 Jan 9;16(1):35. doi: 10.1186/s13018-020-02192-6. PMID 33422084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants previously recruited & enrolled in the post-market approval (PMA) were considered enrolled in this post-approval study (PAS). Additional consent was not required (reviewed and approved by study sites' ethic committees) because the participants had existing consent from the PMA agreeing to be followed to the 10-year postoperative interval necessary for this PAS.
Groups:
- Post Approval Study: Participants implanted with the R3 delta Ceramic Acetabular System (DoD) in the pivotal study.
Period: Overall Study
Arm/Group | Post Approval Study
Started | 135
Completed | 118
Not Completed | 17
Not completed — Death | 7
Not completed — Failures (revision required) | 2
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | Post Approval Study
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Belgium | 61
  Finland | 32
  United Kingdom | 22
  Spain | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (4.73)

OUTCOME MEASURES:

1. Primary Outcome: Implant Survivorship
Description: Number of participants hip implant survivorship with implant survival defined as no revision through 10 years (i.e., 'Hip Survived' or 'Hip Did Not Survive').
Time Frame: 10 Years
Population: Participants with any data available at the time frame specified
Measure: Count of Participants; unit: Participants
Arm/Group | Post Approval Study
Number analyzed (Participants) | 135
Participants
  Hip Survived | 133
  Hip Did Not Survive (Revision Required) | 2

2. Secondary Outcome: Modified Harris Hip Score (mHHS)
Description: The mHHS scoring assessment ranges from 0 (worst) to 100 (best). Scores assessed during the pre-operative, 3-year, 5-year, 7-year and 10-year visit.
Time Frame: Pre-operative, 3-years, 5-years, 7-years, 10-years
Population: Participants with data available at time frames specifies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post Approval Study
Number analyzed (Participants) | 128
score on a scale
  Pre-operative | 47.9 (12.02)
  3-year: number analyzed (Participants) | 111
  3-year | 92 (11.42)
  5-year: number analyzed (Participants) | 106
  5-year | 92.5 (10.61)
  7-year: number analyzed (Participants) | 99
  7-year | 92 (10.83)
  10-year: number analyzed (Participants) | 103
  10-year | 92.6 (9.29)

3. Secondary Outcome: Number of Participants With Radiographic Success
Description: Count of participants with radiographic success, where success is defined as:
  * No radiolucencies greater than 2 mm in 50% or more in any of the cup or stem zones; and
  * No femoral or acetabular subsidence greater than or equal to 5mm from baseline; and
  * No acetabular cup inclination changes greater than 4 degrees (4°)
  Participants who did not meet criteria specified above were considered radiographic failures
Time Frame: 3-years, 5-years, 7-years 10-years
Population: Number of participants with any data available for the time frame specified
Measure: Count of Participants; unit: Participants
Arm/Group | Post Approval Study
Number analyzed (Participants) | 115
Participants
  3-years: Success | 111
  3-years: Failures | 4
  5-years: number analyzed (Participants) | 106
  5-years: Success | 101
  5-years: Failures | 5
  7-years: number analyzed (Participants) | 95
  7-years: Success | 90
  7-years: Failures | 5
  10-years: number analyzed (Participants) | 102
  10-years: Success | 97
  10-years: Failures | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following implantation of the R3 delta Ceramic Acetabular System (DoD) through 10 years.
Description: All adverse events (AE), regardless of their relationship to the study device were included in the safety analyses. Total participants at risk for each adverse event type (i.e., All Cause Mortality, Serious, and Other) indicates those with available AE data collected.
Arm/Group | Post Approval Study
All-Cause Mortality (participants affected / at risk) | 7/135
Serious Adverse Events (participants affected / at risk) | 83/135
Other Adverse Events (participants affected / at risk) | 99/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Approval Study (N=135)
Aseptic implant (acetabular cup) loosening right hip (Product Issues) | 1 (1) — Related to device
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Cervix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Goiter adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — Unrelated
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Unrelated
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Basal cel carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Mesothelium cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Bronchus/lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Unrelated
Rectal/colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Unrelated
Artery sclerosis (Cardiac disorders) | 5 (5) — Unrelated
Cardiac arrhytmia (Cardiac disorders) | 8 (8) — Unrelated
Cerebrovascular infarction (Cardiac disorders) | 4 (4) — Unrelated
Deep vein trombosis (Cardiac disorders) | 2 (2) — Unrelated
Congestive heart failure descompensation (Cardiac disorders) | 3 (3) — Unrelated
Hypertension (Cardiac disorders) | 2 (2) — Unrelated
Insufficienty mitral valve (Cardiac disorders) | 1 (1) — Unrelated
Takotsubo cardiomyopathy (Cardiac disorders) | 1 (1) — Unrelated
TIA (Cardiac disorders) | 1 (1) — Unrelated
Stroke (Cardiac disorders) | 2 (2) — Unrelated
Death (General disorders) | 2 (2) — Unrelated
Abcess (Gastrointestinal disorders) | 2 (2) — Unrelated
Appendicitis (Gastrointestinal disorders) | 2 (2) — Unrelated
Cholecystitis (Gastrointestinal disorders) | 1 (1) — Unrelated
Diarrhea (Gastrointestinal disorders) | 2 (2) — Unrelated
Diverticulosis (Gastrointestinal disorders) | 3 (3) — Unrelated
Fistel (Gastrointestinal disorders) | 2 (2) — Unrelated
Gastro-intestinal bleeding (Gastrointestinal disorders) | 1 (2) — Unrelated
Hernia Inguinalis (Gastrointestinal disorders) | 3 (3) — Unrelated
Rectosigmoidoal polyp (Gastrointestinal disorders) | 1 (1) — Unrelated
Stomach perforation (Gastrointestinal disorders) | 1 (1) — Unrelated
Abdominal pain due to dehydration (Endocrine disorders) | 1 (1) — Unrelated
Diabetes (Endocrine disorders) | 2 (2) — Unrelated
Acute liver failure (Endocrine disorders) | 1 (1) — Unrelated
Multinodular goiter (Endocrine disorders) | 1 (1) — Unrelated
Liver cirrosis (Endocrine disorders) | 1 (1) — Unrelated
Pancreatitis (Endocrine disorders) | 1 (1) — Unrelated
Blepharochalasis (Eye disorders) | 1 (1) — Unrelated
Cataract (Eye disorders) | 10 (15) — Unrelated
Degeneration (Eye disorders) | 2 (2) — Unrelated
Subluxation eye lens (Eye disorders) | 2 (2) — Unrelated
Hypokaliemia (Immune system disorders) | 1 (1) — Unrelated
Surgical wound infection (Infections and infestations) | 1 (1) — Unrelated
Sepsis (Infections and infestations) | 1 (1) — Unrelated
Induced coma due to road traffic accident (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Pelvic fracture due to a fall (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Wound head due to a fall (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Wound in face (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Related to device
Alzheimer (Psychiatric disorders) | 1 (1) — Unrelated
Depression (Psychiatric disorders) | 1 (1) — Unrelated
Stress (extreme) (Psychiatric disorders) | 1 (1) — Unrelated
Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Achilles tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Meniscus tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Muscle tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Disc prolapse (Nervous system disorders) | 1 (1) — Unrelated
Carpal tunnel syndrome right (Nervous system disorders) | 1 (1) — Unrelated
Commotio cerebri (Nervous system disorders) | 2 (2) — Unrelated
Leuco-encefalopathy (Nervous system disorders) | 1 (1) — Unrelated
Corticosubcorticale atrophy (Nervous system disorders) | 1 (1) — Unrelated
Polyneuropathy (Nervous system disorders) | 1 (1) — Unrelated
Pain left hip due to a fall (General disorders) | 1 (1) — Unrelated
Worsening of the polyethylene liner wear + hip left side (General disorders) | 1 (1) — Unrelated
Hysterocele (Reproductive system and breast disorders) | 1 (1) — Unrelated
Benigne prostate hypertrophy (Reproductive system and breast disorders) | 1 (1) — Unrelated
Epidydimitis (Reproductive system and breast disorders) | 1 (1) — Unrelated
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Unrelated
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) — Unrelated
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Unrelated
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Lung oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Pleura fluid (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Lung embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Respiratory sepsis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Respiratory insuficience (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Acetabular component loosening (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Arthrosis (Musculoskeletal and connective tissue disorders) | 5 (6) — Unrelated
broken tooth (General disorders) | 1 (1) — Unrelated
Fracture (Musculoskeletal and connective tissue disorders) | 8 (9) — Unrelated
Contusio (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Foot Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hernia (Musculoskeletal and connective tissue disorders) | 5 (5) — Unrelated
Impingement (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Labral tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Pain (Musculoskeletal and connective tissue disorders) | 4 (4) — Unrelated
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (3) — Unrelated
Revision surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Wound (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Ingrown toenail (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Laceration (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Correction abdominal wall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Headache, right eye visual symptoms for unknown reason (General disorders) | 2 (2) — Unrelated
Hiccup (General disorders) | 1 (1) — Unrelated
Acute Kidney failure (Renal and urinary disorders) | 4 (4) — Unrelated
Hydro-uretronetrosis (Renal and urinary disorders) | 1 (1) — Unrelated
Hematurie (Renal and urinary disorders) | 2 (2) — Unrelated
Chronic Kidney failure (Renal and urinary disorders) | 1 (1) — Unrelated
Hydrometrose (Renal and urinary disorders) | 1 (1) — Unrelated
Renal insufficiency (Renal and urinary disorders) | 2 (2) — Unrelated
Subnephrotic proteinaria due to her nephropathy (Renal and urinary disorders) | 1 (1) — Unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Approval Study (N=135)
Hypertension (Vascular disorders) | 2 (2) — Unrelated
Claudication (Vascular disorders) | 1 (1) — Unrelated
Diverticulitis aorta (Vascular disorders) | 1 (1) — Unrelated
Chronic venous insufficiency (Vascular disorders) | 3 (3) — Unrelated
Syncope (Vascular disorders) | 1 (1) — Unrelated
Aneurysma (Vascular disorders) | 1 (1) — Unrelated
AV-block Grade I (Vascular disorders) | 1 (1) — Unrelated
Artery sclerosis (Vascular disorders) | 2 (2) — Unrelated
Cardiac arrhytmia (Vascular disorders) | 2 (2) — Unrelated
Deep vein trombosis (Vascular disorders) | 1 (1) — Unrelated
Sinnus of arterial insufficiency (Vascular disorders) | 1 (1) — Unrelated
Peripheral arterial disease (Vascular disorders) | 1 (1) — Unrelated
Headache (Vascular disorders) | 1 (1) — Unrelated
Multiple brain ischemia chronic (Vascular disorders) | 1 (1) — Unrelated
Abdominal pain (Gastrointestinal disorders) | 2 (2) — Unrelated
Hemorrhagia Ex Ano (Gastrointestinal disorders) | 2 (2) — Unrelated
Fecal incontinence (Gastrointestinal disorders) | 1 (1) — Unrelated
Diverticulitis (Gastrointestinal disorders) | 2 (2) — Unrelated
Nausea (Gastrointestinal disorders) | 2 (2) — Unrelated
Hemorrhoids (Gastrointestinal disorders) | 1 (1) — Unrelated
Anal swelling (Gastrointestinal disorders) | 1 (1) — Unrelated
Pyrosis (Gastrointestinal disorders) | 1 (1) — Unrelated
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — Unrelated
Gastric pain (Gastrointestinal disorders) | 1 (1) — Unrelated
Tinnitus (Ear and labyrinth disorders) | 1 (1) — Unrelated
Otitis externa (Ear and labyrinth disorders) | 1 (1) — Unrelated
Hearing impairment (Ear and labyrinth disorders) | 4 (4) — Unrelated
Vertigo (Ear and labyrinth disorders) | 3 (3) — Unrelated
Tube dysfunction (Ear and labyrinth disorders) | 1 (1) — Unrelated
Cholelithiasis (Endocrine disorders) | 2 (2) — Unrelated
Hypovitaminosis (Endocrine disorders) | 1 (1) — Unrelated
Gout (Endocrine disorders) | 2 (2) — Unrelated
Liver steatosis (Endocrine disorders) | 2 (2) — Unrelated
Hypercholesterolemia (Endocrine disorders) | 2 (2) — Unrelated
Cholecystalithiosis (Endocrine disorders) | 1 (1) — Unrelated
Enlarged thyroid gland (Endocrine disorders) | 1 (1) — Unrelated
Cataract (Eye disorders) | 4 (4) — Unrelated
Retinal rupture (Eye disorders) | 1 (1) — Unrelated
PCO (Eye disorders) | 1 (1) — Unrelated
Groin pain due to tendinopathy (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Deteriorating pain in groin right hip (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Slightly higher CRP (Immune system disorders) | 1 (1) — Unrelated
Rheuma (Immune system disorders) | 1 (1) — Unrelated
Heterotopic ossification of hip seen on xray (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Peri-articular ossification (Musculoskeletal and connective tissue disorders) | 6 (6) — Unrelated
Worsening of peri-articular ossification (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Discomfort lateral aspect hip (General disorders) | 2 (2) — Device related
Occasional mild discomfort in groin and hip (General disorders) | 1 (1) — Device related
Cellulitis (Infections and infestations) | 1 (1) — Unrelated
Herpes (Infections and infestations) | 2 (2) — Unrelated
Infection surgical wound (Infections and infestations) | 1 (1) — Unrelated
Flu (Infections and infestations) | 2 (2) — Unrelated
Patient fell down (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Allergic reaction (food) (Injury, poisoning and procedural complications) | 1 (1) — Unrelated
Dementia (Psychiatric disorders) | 2 (2) — Unrelated
Depression (Psychiatric disorders) | 1 (1) — Unrelated
Memory decline (Psychiatric disorders) | 1 (1) — Unrelated
Anxiety (Psychiatric disorders) | 1 (1) — Unrelated
Oedema legs (Blood and lymphatic system disorders) | 1 (1) — Unrelated
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Chondrocalcinosis menisci (Musculoskeletal and connective tissue disorders) | 1 (2) — Unrelated
Elastofibroma (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Inflammation bursa iliopsoas (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Fibrostosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Impingement (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Infection tendon (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
muscular reumatism (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Muscle tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Menisci tears (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Rupture tendon (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Symphysitis of pubis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Tendinopathy (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Tendinosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Tendostosis (Musculoskeletal and connective tissue disorders) | 2 (3) — Unrelated
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Tennis elbow (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Trochanteritis (Musculoskeletal and connective tissue disorders) | 3 (3) — Unrelated
Radicular pain in lower extremity (Ischias) (Nervous system disorders) | 2 (2) — Unrelated
Sleep apnea (Nervous system disorders) | 2 (2) — Unrelated
Neuropatic pain (Nervous system disorders) | 1 (1) — Unrelated
Horner syndrome (Nervous system disorders) | 1 (1) — Unrelated
Dizziness cervical origin (Nervous system disorders) | 1 (1) — Unrelated
Unexplained bruising on lower left calf (General disorders) | 1 (1) — Unrelated
Afonia (General disorders) | 1 (1) — Unrelated
Fever and color wound right leg (General disorders) | 1 (1) — Unrelated
Fever (General disorders) | 1 (1) — Unrelated
Unexplained pain of operated hip (General disorders) | 1 (1) — Device related
Pain (General disorders) | 1 (1) — Device related
Iliopsoas bursitis (General disorders) | 1 (1) — Device related
Pain (General disorders) | 2 (2) — Unrelated
Chest pain (General disorders) | 2 (2) — Unrelated
Headache (General disorders) | 4 (5) — Unrelated
Pain in hip (General disorders) | 1 (1) — Unrelated
Breast pain (General disorders) | 1 (1) — Unrelated
Adverse reaction to metal debris (Product Issues) | 1 (1) — Device related
Prostatitis (Reproductive system and breast disorders) | 1 (1) — Unrelated
Benigne prostate hypertrophy (Reproductive system and breast disorders) | 1 (1) — Unrelated
Epydimitis left testes (Reproductive system and breast disorders) | 1 (1) — Unrelated
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Unrelated
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Unrelated
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Unrelated
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Arthrosis (Musculoskeletal and connective tissue disorders) | 19 (28) — Unrelated
Capsular irritation around left hip and groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Cervicalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Cervicobrachialgie (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Chondromalacie (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Contusion (Musculoskeletal and connective tissue disorders) | 9 (9) — Unrelated
Discopathy (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Dupuytren dig 5 right hand (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) — Unrelated
Hallux rigidus (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Hallux Valgus (Musculoskeletal and connective tissue disorders) | 2 (3) — Unrelated
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) — Unrelated
Heel spur (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Lumbalgie (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) — Unrelated
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Painful metatarsophalangeal joint (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Pain in hip (Musculoskeletal and connective tissue disorders) | 4 (4) — Unrelated
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Pain in foot (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Peri-articular ossification (Musculoskeletal and connective tissue disorders) | 3 (3) — Unrelated
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Pins and needles left leg (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 (5) — Unrelated
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) — Unrelated
Cervical vertebrae stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Trochanteritis (Musculoskeletal and connective tissue disorders) | 2 (2) — Unrelated
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Active keratosis (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Solar Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated
Dermatochalasis (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated
Exostosis in the heel (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Wound on left hip - along previous surgery wound (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Wound right knee and lower leg due to a fall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Erythema due to bites of insects (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Removal birthmark nose (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Skin tear left arm due to a fall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Cut left little finger (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Panniculitis right knee (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Wound left index finger (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Subunguaal hematoma right finger (3) (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Wound nose due to a fall (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Seborrheic keratosis irritation (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Keratosis actinica (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated
Prolonged chest pain (General disorders) | 1 (1) — Unrelated
Intermittent flare ups of neck pain and right arm pain (General disorders) | 1 (1) — Unrelated
Slight stiffness in right hip (Musculoskeletal and connective tissue disorders) | 1 (1) — Device related
Benigne paroxysmale positionings vertigo (BPPV) (Ear and labyrinth disorders) | 1 (1) — Unrelated
Trochanteritis right hip (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Urinary tract infection (Renal and urinary disorders) | 3 (4) — Unrelated
Cystitis acute (Renal and urinary disorders) | 1 (1) — Unrelated
Ovarium cyste (Renal and urinary disorders) | 1 (1) — Unrelated
Prostate hypertrophy (Renal and urinary disorders) | 3 (3) — Unrelated
Haematuria (asymptomatic) (Renal and urinary disorders) | 1 (1) — Unrelated
Benign tumor tonsilla (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Rectal/colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated
Meningeoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated

LIMITATIONS AND CAVEATS:
At the 10+ Year interval, the follow-up rates that require collection of additional data for the secondary endpoints, ActualA-In-Window and ActualA, are 77.0% and 78.6%, respectively, for all hips. The additional analyses that were done to assess the impact of protocol deviations incurred including those resulting from the COVID-19 pandemic support that the missing data are unlikely to have an impact on the primary or secondary endpoint results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03566082/Prot_SAP_000.pdf